CLINICAL TRIAL: NCT05317962
Title: Cardiac Manifestations of COVID-19 in Patients Admitted to Hospital
Brief Title: COVID-19 Echo Study
Status: Completed | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRC/2020/002
Record Dates: First submitted 2020-09-09; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2020-04

CONDITIONS: Covid-19; Cardiac Disease
Keywords: Echocardiography
MeSH Terms: conditions — COVID-19; Heart Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive patients admitted to hospital
  Interventions: Diagnostic Test: Transthoracic echocardiogram

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiogram — Abbreviated transthoracic echocardiogram

SUMMARY:
Investigation of the cardiac manifestations of COVID-19 in patients admitted to hospital

DETAILED DESCRIPTION:
The COVID-19 disease (caused by SARS-CoV-2) predominantly affects the lungs causing a pneumonia which can become severe and lead to death via a severe inflammatory response in the lungs for which patients require admission to intensive care units (ICU) and artificial ventilation of their lungs. However, early reports from China have documented an element of injury to the heart present in up to 20% of patients. They have also documented patients who have died on ICU from heart injury rather than lung injury in COVID-19 positive patients. There are increasing numbers of reports of patients with COVID-19 having significant inflammation of the heart. What is not known is the prevalence of significant inflammation of the heart secondary to the SARS-CoV-2 and also what the significance of the injury to the heart shown in 20% of patients through blood tests really represents. That is to say is the injury significant to the outcome of the patient?

In order to investigate this, it is proposed to conduct a heart scan in COVID-19 positive patients in hospital to determine what form of heart injury is caused by the disease as well as determining it's prevalence and whether a heart scan helps in risk stratifying the patient in terms of outcome. If it is found that there is a significant amount of heart injury done by the SARS-CoV-2 and it can be determined this at an early stage with a heart scan it may be possible to start a more aggressive strategy for the patient's management in hospital to reduce the chance of death. Alternatively, if it is found that the incidence of heart injury is low and a heart scan makes no difference to the management of the patient, medical teams can be advised of this.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Positive swab or serology for COVID-19
3. Referred for echocardiographic evaluation for clinical reasons
4. Willing and able to give assent

Exclusion Criteria:

1. Known hypersensitivity to perflutren or known excipients in LUMINITY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the cardiology department at Northwick Park Hospital to have a transthoracic echocardiogram who have also tested positive for COVID-19,
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiac abnormalities and relationship to admission to ICU | 6 weeks from start of admission

SECONDARY OUTCOMES:
Prevalence of cardiac abnormalities and relationship to need for mechanical ventilation | 6 weeks from start of admission
Prevalence of cardiac abnormalities and relationship to death or discharge | 6 weeks from start of admission

CONTACTS AND LOCATIONS:
Overall Officials: Prof Roxy Senior, MD, Principal Investigator — North West London University Healthcare NHS Trust
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No